CLINICAL TRIAL: NCT05508555
Title: Effect of Intraoperative Hyperthermic Intrathoracic Chemotherapy After Pleurectomy Decortication for Treatment of Malignant Pleural Mesothelioma.
Brief Title: Effect of HITHOC After Pleurectomy Decortication for Treatment of Malignant Pleural Mesothelioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HITHOC after PD in MPM
Record Dates: First submitted 2022-08-01; First posted 2022-08-19 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Malignant Pleural Mesothelioma; Chemotherapy Effect
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HITHOC group (Active Comparator): the group that will receive HITHOC after pleurectomy decortication
  Interventions: Procedure: hyperthermic intrathoracic chemotherapy
- pleurectomy decortication without HITOC (No Intervention): the group who received pleurectomy decortication without HITHOC

INTERVENTIONS:
Procedure: hyperthermic intrathoracic chemotherapy — application of chemotherapeutic agent intrathoracic under hyperthermic conditions
  Arms: HITHOC group

SUMMARY:
Malignant pleural mesothelioma (MPM) is an aggressive malignancy of the pleural lining with exceptionally poor survival. Median survival from diagnosis is less than 12 months (1). The widespread use of asbestos in past decades together with the long latency of MPM are responsible for the still increasing incidence of MPM (2), affecting 7-40 people per million inhabitants depending on the geographic region (3). The main therapeutic strategies for MPM are surgery, chemotherapy, and radiation therapy (RT). Multimodality treatment for MPM is a topic that has been attracting a lot of attention from researchers, as therapeutic modalities such as surgery, chemotherapy, or radiotherapy have not proven to be effective as single-modality treatments (4). surgery alone is not able to achieve microscopic complete (R0) resection. Therefore, combined treatment modalities have been established in many centres during the last years to achieve a better local tumor control with increasing overall survival (5). In this regard, hyperthermic intrathoracic or intrapleural chemotherapy has been used as one of the multimodality therapies. Intrapleural injection of cytotoxic drugs with hyperthermic perfusion has been proved to enhance cytotoxic effect on tumor cells with limited systemic side effect (6). While cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy (HIPEC) has become a standard therapy for intraperitoneal original carcinoma or carcinomatosis peritonei such as pseudomyxoma and colorectal cancer induced ascites (7), limited studies have been reported on the application of hyperthermic intrathoracic chemotherapy (HITHOC) in combination with cytoreductive surgery for the treatment of the malignant pleural mesothelioma (8). With the application of the HITOC after macroscopic complete pleural tumour resection, it is expected to obtain better local tumour control, and thereby improve progression-free as well as overall survival (9).

In this study, we aim to compare results of HITHOC after P/D versus P/D alone in managing patients with localised MPM and our main outcomes are disease free survival, overall survival and possible perioperative complications.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a fatal malignancy with limited options of therapies including surgery, radiotherapy and chemotherapy (10). extensive tumor extraction can be achieved with either extrapleural pneumonectomy (EPP) or extended pleurectomy/decortication (P/D. However, significant proportion of patients have relapse of the disease following EPP or P/D and they usually die within a few months (11). Thus, surgery-based multimodality therapies have been clinically explored in the past decades. Intraoperative intrapleural injection of cytotoxic drugs, such as cisplatin, doxorubicin, gemcitabine, or epirubicin, with hyperthermic perfusion at the time of surgery, i.e, hyperthermic intrathoracic chemotherapy (HITHOC), is a widely used method of multimodality treatment for MPM to optimize local disease control (12). The most popular cytotoxic drugs used for HITHOC were cisplatin followed by doxorubicin and mitomycin C, and 41-43 ◦C was most commonly used in HITHOC. The standard time for infusion was 60-90 min across the studies. Intrathoracic instillation of chemotherapeutic agents allows for a much higher concentration of the drug in the pleural cavity potentially improving the cytotoxic effect to the tumor cells and minimizing systemic adverse effects (13).

ELIGIBILITY:
Inclusion Criteria:

* patients presented with localised MPM are the main target and histopathological diagnosis of MPM is made via video-assisted thoracoscopic surgery or open multiple pleural biopsies.

Exclusion Criteria:

* patients with stage III or IV MPM in which cytoreductive surgery has no role.
* Patients underwent extrapleural pneumonectomy (EPP) as a cytoreductive surgery , because we are focusing on P/D only either conventional P/D or extended P/D

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
disease free survival or time to recurrence | Through out the whole study with maximum of 2 years
  time from clearance of disease till onset of recurrence of same disease
overall survival | till mortality of the case or 2 years maximum
  survival of the cases till mortality

SECONDARY OUTCOMES:
comorbidities | Through out the whole study duration with maximum of two years
  complications that may encounter either pre , intra or post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hany Hassan El sayed, prof Dr., Study Director — hanyhassan77@hotmail.com
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

REFERENCES:
- [Background] Cao C, Tian D, Park J, Allan J, Pataky KA, Yan TD. A systematic review and meta-analysis of surgical treatments for malignant pleural mesothelioma. Lung Cancer. 2014 Feb;83(2):240-5. doi: 10.1016/j.lungcan.2013.11.026. Epub 2013 Dec 6. PMID 24360321
- [Background] Opitz I. Management of malignant pleural mesothelioma-The European experience. J Thorac Dis. 2014 May;6 Suppl 2(Suppl 2):S238-52. doi: 10.3978/j.issn.2072-1439.2014.05.03. PMID 24868442
- [Background] Friedberg JS, Simone CB 2nd, Culligan MJ, Barsky AR, Doucette A, McNulty S, Hahn SM, Alley E, Sterman DH, Glatstein E, Cengel KA. Extended Pleurectomy-Decortication-Based Treatment for Advanced Stage Epithelial Mesothelioma Yielding a Median Survival of Nearly Three Years. Ann Thorac Surg. 2017 Mar;103(3):912-919. doi: 10.1016/j.athoracsur.2016.08.071. Epub 2016 Nov 5. PMID 27825687
- [Background] Maziak DE, Gagliardi A, Haynes AE, Mackay JA, Evans WK; Cancer Care Ontario Program in Evidence-based Care Lung Cancer Disease Site Group. Surgical management of malignant pleural mesothelioma: a systematic review and evidence summary. Lung Cancer. 2005 May;48(2):157-69. doi: 10.1016/j.lungcan.2004.11.003. Epub 2005 Jan 5. PMID 15829316